CLINICAL TRIAL: NCT02073591
Title: A Phase IV, Open Label, Single Arm, Multicenter, Observational Study to Evaluate the Correlation Between PEST and SCORAD Score in the Management of Atopic Dermatitis With Use of Ceradan® Regimen in Children Aged Six Months to Six Years
Brief Title: Correlation Study Between PEST and SCORAD in Management of Atopic Dermatitis With Ceradan® Regimen
Acronym: COPES
Status: Completed | Type: Observational
Sponsor: Hyphens Pharma Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: HYP2013/001
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Atopic Dermatitis
Keywords: Children; Atopic Dermatitis; Ceradan; PEST; SCORAD
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ceradan Regimen: Ceradan Cream and Ceradan Wash
  Interventions: Other: Ceradan Cream; Other: Ceradan Wash

INTERVENTIONS:
Other: Ceradan Cream
Other: Ceradan Wash

SUMMARY:
This is a prospective, open label, single arm, and observational and multicenter study to assess the correlation between PEST and SCORAD scores in the management of AD with the Ceradan® regimen.

DETAILED DESCRIPTION:
All eligible patients shall apply permitted topical steroid(s) according to standard local practice

For the entire study period, patients should apply Ceradan Cream® liberally twice daily or more, if required and use a non-soap based wash once or twice daily.

At the screening visit, patients will receive a diary card and will be asked to track their atopic dermatitis symptoms for 12 weeks.

Retrospective information on other topical treatments used will be collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged ≥6 months to ≤6 years
* Baseline PEST score of 3- 4
* Diagnosis of mild to moderate atopic dermatitis, with grading of 3 to11, as per the NESS
* Diagnosis of current flare (increased dryness, itching, redness, swelling and general irritability) at baseline visit according to Investigator's judgement
* Patients who have not visited the dermatologist before (dermatologist-naïve)
* Agree to participate and provide written consent by parent or guardian (and assent if applicable)

Exclusion Criteria:

* History of severe episodes of atopic dermatitis (for example: oozing, crusts)
* Clinical signs of skin infection (viral, bacterial or fungal)
* Grading of >11 as defined by the Nottingham Eczema Severity Score (NESS) within 3 months prior to study inclusion
* Known reaction or allergy to test drug or excipients or steroids
* History of cutaneous or systemic viral (including HIV or AIDS), cutaneous mycotic or cutaneous bacterial disease requiring a topical or systemic therapy during the study period
* Patients who are receiving any investigational drug or who have taken part in a clinical study with an investigational drug within three months prior to the start of study treatment
* The patient has been exposed to below therapy within the set timeframe:

  i. Systemic administration of corticosteroid - four weeks; ii. Systemic administration of immunosuppressive drugs - four weeks; iii. UV therapy four weeks
* Any serious medical condition which, in the opinion of the investigator, may interfere with the evaluation of the results
* Parents/guardians may be unable to complete the patient diaries or questionnaires

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children Aged Six Months to Six Years with Atopic Dermatitis
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Correlation between the mean Patient Eczema Severity Time (PEST) score and mean Scoring Atopic Dermatitis (SCORAD) Index at Week 4 and Week 12, as compared to baseline | 12 weeks
  Correlation will be assessed by Pearson correlation at baseline, Week 4 and Week 12 between both scores. Karl Pearson correlation coefficient (ρ) will be provided. Percent Change from Baseline will be calculated for Week 4 and Week 12 and correlation will also be calculated for it.

SECONDARY OUTCOMES:
Efficacy by change in SCORAD score at Week 4 and Week 12 as compared to baseline | 12 weeks
Efficacy by change in AUC PEST score at Week 4, Week 12 as compared to baseline and three months prior to baseline | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - National Skin Centre, Singapore

REFERENCES:
- [Derived] Koh MJ, Giam YC, Liew HM, Foong AY, Chong JH, Wong SMY, Tang MBY, Ho MSL, Tan LS, Mason JM, Cork MJ. Comparison of the Simple Patient-Centric Atopic Dermatitis Scoring System PEST with SCORAD in Young Children Using a Ceramide Dominant Therapeutic Moisturizer. Dermatol Ther (Heidelb). 2017 Sep;7(3):383-393. doi: 10.1007/s13555-017-0186-1. Epub 2017 Jun 14. PMID 28616853